CLINICAL TRIAL: NCT06920342
Title: Investigating Attitudes to Gynaecological Rapid Access, Cancer Exclusion and Follow Up Location (GRACEFUL Study)
Brief Title: Attitudes to Gynae Oncology Care Location - GRACEFUL
Acronym: GRACEFUL
Status: Recruiting | Type: Observational
Sponsor: Somerset NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 339158
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic Cancers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Gynaecological oncology (cancer) place of care is often based on evolution of services, along historical professional boundaries, rather than user needs or preferences. The investigators aim to gather views of patients in the United Kingdom (UK) on their preferred place of care for investigation, treatment and follow-up of gynaecological cancer. An initial scoping review found no previous work in this area. Pilot work, performed to inform local re-organisation of services, found that 53% of participants were somewhat or very unhappy to have care co-located with O&G services. Specifically, two key themes were identified through content analysis of free-text comments: "environment and getting this right is vital"; and "our cancer should be the priority".

However, via a BGCS survey, the investigator found that healthcare professionals (HCPs) underestimated strong patient preferences. Of those who see patients within O&G services, only 50% said patients were seen at separate times/locations from obstetric patients. The investigators want to expand on these pilot data to better understand how to design services that better meet our patients' needs. The investigators will conduct a survey to ascertain service users' attitudes to location of services, collecting quantitative data & qualitative data, including opportunities for feedback in free text. The investigator will conduct analysis using standard statistical methods & content analysis of free-text responses. Submissions will be anonymous & no identifiable data will be collected routinely, unless volunteered by the respondent. The investigator will ask a subset of ~30 participants to undertake a telephone/virtual-based semi-structured interview to further explore understanding on attitudes to location of care more generally. A topic guide will be developed, informed by the Theoretical Framework of Acceptability. Interviews will be audio-recorded with consent, transcribed verbatim & anonymised. The anonymised transcripts will be analysed using a form of Thematic Analysis. These findings should help to shape future health care service sensitive to patient need.

ELIGIBILITY:
Inclusion Criteria:

- Female Aged 18 or over Able to give informed consent Have been referred to secondary care with a suspected gynaecological cancer, or have previously been diagnosed with a gynaecological malignancy

Exclusion Criteria:

- Male Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — non
Study Population: UK
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-02-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
Graceful 1 | 5 years
  Patient-reported outcomes of acceptability of different clinic co-locations and the impact of different services.

CONTACTS AND LOCATIONS:
Locations (1):
- Somerset NHS Foundation Trust, Taunton, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No